CLINICAL TRIAL: NCT02169492
Title: Evaluation of the ReVive SE Device for Intra-Arterial Thrombectomy in Acute Ischemic Stroke: An Observational, Prospective and Multicenter Study
Brief Title: Evaluation of the ReVive SE Device for Intra-Arterial Thrombectomy in Acute Ischemic Stroke
Acronym: Re-ACT
Status: Completed | Type: Observational
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Other Study IDs: NV-PMK-1203
Record Dates: First submitted 2014-06-13; First posted 2014-06-23 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Stroke
Keywords: Thrombectomy; Stroke; ReVive SE
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the ReVive SE (Self- Expanding) Neurothrombectomy Device in subjects requiring mechanical thrombectomy when used according to its Instruction for use (IFU).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Clinical signs consistent with acute ischemic stroke
3. No pre-stroke functional dependence (pre-stroke Modified Rankin Score ≤ 1)
4. NIHSS ≥ 6,, assessed within two hours before treatment with ReVive SE
5. Large (≥ 1.5mm) and proximal vessel occlusion (presenting TICI score of 0 or 1) of MCA (M1-M2), dICA, or BA confirmed by CT/MR angiography that it is accessible to the ReVive SE.
6. Treatment initiated within 8 hours after symptom onset (first ReVive SE pass made within 6 hours
7. Subject or legally authorized representative has provided informed consent on data collection, and consent is documented

Exclusion Criteria:

1. Life expectancy of less than 90 days
2. Neurological signs that are rapidly improving prior to or at time of treatment (NIHSS improves at least 4 points between subject presentation and treatment initiation)
3. Subject is either exhibiting clinical signs suggestive of, or there is angiographic evidence of bilateral stroke
4. Prior use of any other mechanical device to treat this stroke (e.g., Merci Retriever, Penumbra, Solitaire, Trevo, Mindframe, Phenox, stent)
5. Known bleeding diathesis:

   1. Current use of oral anticoagulants (eg, warfarin sodium) with International Normalized Ratio (INR) > 3;
   2. Administration of heparin or Novel Oral AntiCoagulants (NOAC, eg Dabigatran, Rivaroxaban) within 48 hours preceding the onset of stroke and have an abnormal activated partial thromboplastin time (aPTT) at presentation; and/or
   3. Platelet count < 100,000/mm3
6. Glucose <50 mg/dL (2.8 mmol, 2.6mM)
7. Uncontrolled hypertension (SBP>185 or DBP>110) refractory to pharmacological management
8. Known hypersensitivity or allergy to nitinol and/or radiographic contrast agents
9. Pregnancy or lactating female
10. Subject already enrolled in a clinical study involving experimental medication or device

    Imaging Exclusion criteria:
11. CT scan or MRI with evidence of acute intracranial hemorrhage, mass effect and/or intracranial tumor.
12. Angiographic evidence of carotid dissection, or high grade stenosis (> 50% stenosis of the artery proximal to the target vessel) that will prevent access to the clot, or cerebral vasculitis
13. Blood vessel with extreme tortuosity or other conditions preventing the access of the device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects requiring mechanical thrombectomy
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale | 90 days
  Functional Independence of subjects as defined by modified Rankin Scale (mRS) ≤2 at 90 days post-procedure.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | 90 days

OTHER OUTCOMES:
emboli occurence | 90
symptomatic intracranial hemorrhage (sICH) | 90 days
Mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hoehn, MD, Study Director — Codman Neuro
Locations (8):
- France (8):
  - CHU Bordeaux, Bordeaux
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU de Colmar, Colmar
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - CHU La Timone, Marseille
  - CHU St Etienne, Saint-Etienne
  - Hôpital Bretonneau, Tours